CLINICAL TRIAL: NCT03555461
Title: Analysis of EPA® (a Food Intake Assessment Tool) as a Screening Test for Malnutrition in General Medicine
Acronym: GEN-EPA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3087-GEN-EPA
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to evaluate the sensitivity of the EPA® for screening for malnutrition in general medicine in adults.

ELIGIBILITY:
Inclusion Criteria:

* To be an adult,
* Consulting the principal investigator, a general practitioner in his activity of substitute doctor,
* During the inclusion period,
* Not opposed to participating in the study.

Exclusion Criteria:

* Patients benefiting from artificial nutrition,
* Patients with advanced dementia,
* Pregnant or postpartum women,
* Patients who do not understand or speak French,
* Patients treated with diuretics who have had a change in treatment dosage during the last 6 months,
* Patients for whom weight measurement is not possible in the office (wheelchair, disability ...),
* Patients who have already been included once,
* Patients who have had surgery for obesity,
* Major persons subject to legal protection (legal safeguards, guardianship, tutorship), persons deprived of their liberty, ...

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting a general practioner in his activity of substitute doctor,
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

PRIMARY OUTCOMES:
presence or absence of malnutrition | The inclusion day
  presence or absence of malnutrition based on BMI and / or percentage of weight loss
Score EPA | The inclusion day
  score obtained with the EPA® tool (assessment of food intake)

CONTACTS AND LOCATIONS:
Overall Officials: Ronan PhD Thibault, Principal Investigator — Rennes University Hospital
Locations (3):
- France (3):
  - Cabinet médical des Rosiers, Acigné
  - Cabinet médical des Docteurs Le Vagueres et Godard,, Berné
  - Cabinet médical du Dr Berthier,, Languidic